CLINICAL TRIAL: NCT06490705
Title: Chang Gung Memorial Hospital At Linkou
Brief Title: The Efficacy of Tongue Exercises on Swallowing Function in the Elderly with Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Medical Foundation (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Kao, Shu-Hua, Chang Gung Memorial Hospital at Linkou, Chang Gung Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChangGungMF
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-06

CONDITIONS: Dysphagia, Oropharyngeal
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: This is a longitudinal research design using cluster randomization. Participants were randomly divided into three groups by computer, 30 people per group:
  Group 1 received tongue resistance exercises. Group 2 received both tongue strengthening exercises and tongue resistance exercises.
  Group 3: control group received oral and cheek bulging exercises. The exercise intervention is divided into two stages. After completing the pre-test (T1), the first stage of 12 weeks of exercise begins, with evaluations conducted at the 4th week (T2), 8th week (T3), and 12th week (T4). After a 12-week rest period (T5), the second phase of Boosters exercise is conducted for another 12 weeks, followed by an immediate post-test (T6) and a final evaluation after another 12 weeks of rest (T7). Participants received exercise 6 days a week, 3 times a day (before meals), with each session lasting 30 minutes.
Who Masked: Participant
Masking Description: The study design uses cluster randomization to assign subjects to three groups different exercise groups. This study employs a single-blind design to minimize bias, where the participants are blinded to the group allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tongue resistance exercises (Experimental): Participants received tongue resistance exercises 6 days a week, 3 times a day (before meals), with each session lasting 30 minutes.
  The exercise intervention is divided into two stages. After completing the pre-test (T1), the first stage of 12 weeks of exercise begins, with evaluations conducted at the 4th week (T2), 8th week (T3), and 12th week (T4). After a 12-week rest period (T5), the second phase of Boosters exercise is conducted for another 12 weeks, followed by an immediate post-test (T6) and a final evaluation after another 12 weeks of rest (T7).
  Interventions: Other: tongue resistance exercises, tongue strengthening exercises and tongue resistance exercises
- Tongue strengthening exercises and tongue resistance exercises (Experimental): Participants received tongue strengthening exercises and tongue resistance exercises 6 days a week, 3 times a day (before meals), with each session lasting 30 minutes.
  The exercise intervention is divided into two stages. After completing the pre-test (T1), the first stage of 12 weeks of exercise begins, with evaluations conducted at the 4th week (T2), 8th week (T3), and 12th week (T4). After a 12-week rest period (T5), the second phase of Boosters exercise is conducted for another 12 weeks, followed by an immediate post-test (T6) and a final evaluation after another 12 weeks of rest (T7).
  Interventions: Other: tongue resistance exercises, tongue strengthening exercises and tongue resistance exercises
- cheek bulging exercises (Active Comparator): Participants received cheek bulging exercises6 days a week, 3 times a day (before meals), with each session lasting 30 minutes.
  The exercise intervention is divided into two stages. After completing the pre-test (T1), the first stage of 12 weeks of exercise begins, with evaluations conducted at the 4th week (T2), 8th week (T3), and 12th week (T4). After a 12-week rest period (T5), the second phase of Boosters exercise is conducted for another 12 weeks, followed by an immediate post-test (T6) and a final evaluation after another 12 weeks of rest (T7).
  Interventions: Other: tongue resistance exercises, tongue strengthening exercises and tongue resistance exercises

INTERVENTIONS:
Other: tongue resistance exercises, tongue strengthening exercises and tongue resistance exercises — 6 days a week, 3 times a day (before meals), with each session lasting 30 minutes. Don't hold your breath during exercise.
  Before conducting the study, all participants received a complete explanation of the purpose, risks, and procedures of the investigation, and provided written informed consent. Procedures were in accordance with the ethical standards of the committee on human experimentation at the institution at which the work was conducted and this study was approved by the Institutional Review Board.
  Other Names: cheek bulging exercises

SUMMARY:
The purpose of this study is to explore the effects of tongue muscle strength and resistance exercises on dysphagia, tongue muscle strength, oral hygiene, repetitive saliva swallowing, nutrition, depression, and swallowing-related quality of life in frail elderly people with mild cognitive impairment in the community.

This is a longitudinal research design using cluster randomization. Participants were randomly divided into three groups by computer: Experimental Group 1 received tongue resistance exercises; Experimental Group 2 received both tongue strengthening exercises and tongue resistance exercises; and the control group received oral and cheek bulging exercises.

DETAILED DESCRIPTION:
Recruitment was carried out in nursing homes, day passport centers, and community care centers in New Taipei City and Taoyuan City, Taiwan. The subjects were elderly people aged 65 years or older with cognitive impairment and frailty, recruited from November 19, 2021, to January 25, 2024.Participants were randomly divided into three groups by computer, 30 people per group, Group 1 received tongue resistance exercises, Group 2 received both tongue strengthening exercises and tongue resistance exercises, Group 3: control group received oral and cheek bulging exercises.

The exercise intervention is divided into two stages. After completing the pre-test (T1), the first stage of 12 weeks of exercise begins, with evaluations conducted at the 4th week (T2), 8th week (T3), and 12th week (T4). After a 12-week rest period (T5), the second phase of Boosters exercise is conducted for another 12 weeks, followed by an immediate post-test (T6) and a final evaluation after another 12 weeks of rest (T7). Participants received exercise 6 days a week, 3 times a day (before meals), with each session lasting 30 minutes.

Before conducting the study, all participants received a complete explanation of the purpose, risks, and procedures of the investigation, and provided written informed consent. Procedures were in accordance with the ethical standards of the committee on human experimentation at the institution where the work was conducted, and this study was approved by the Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* A. Elderly individuals aged 65 years and above.
* B. Frailty assessment in older adults: Score of at least 1 point.
* C. Cognitive function assessment: Score of >=16 for individuals with no education; >=20 for those with elementary education; >=24 for those with junior high school education or higher.

Exclusion Criteria:

* A. Severe communication barrier.
* B. Unable to move independently or requires assistance.
* C. Unable to raise head or neck.
* D. Recent use of anticholinergic medications, asthma medications, or central nervous system depressants (Benzodiazepines).
* E. Aspiration pneumonia.
* F. Tracheostomy in place.
* G. Neuromuscular disorder.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Frailty assessment | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  Based on the Fried 2001 frailty assessment scale, there are 5 items. The assessment takes only 3 minutes and uses a scoring system of 0 and 1. The possible total score ranges from 0 to 5 points, with higher scores indicating a more severe tendency towards frailty.
Activities of Daily Living (ADL) | OT1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Activities of Daily Living (ADL) Assessment Scale consists of 10 items: eating, transferring, personal hygiene, toileting, bathing, walking on flat ground, climbing stairs, dressing and undressing, bowel control, and bladder control. Each item is graded on a scale of 2-4, ranging from complete dependence to complete independence, with scores incrementing by 5 points. The total score is out of 100 points. Scores from 0 to 20 indicate complete dependence; scores from 21 to 60 indicate severe dependence; scores from 61 to 90 indicate moderate dependence.
Instrumental Activities of Daily Living (IADLs) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Instrumental Activities of Daily Living (IADL) Assessment consists of 8 items, each scored dichotomously (1 or 0), with a maximum total score of 8 points. The number of lost functions helps differentiate the severity of functional impairment, with higher scores indicating greater independence in older adults. The assessment is based on performance over the past month, obtained through observation, interviews with the individual, caregivers, or institutional records. The maximum score is 8 points; for male subjects, cooking, laundry, and housekeeping are not assessed, reducing the total score to 5 points. Mild disability is defined as needing assistance in three or more of the following five areas: shopping, going out, cooking, housekeeping, and laundry.
Mini-Mental State Examination (MMSE) | Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Mini-Mental State Examination (MMSE) evaluates cognitive functions across five domains: orientation, registration, attention and calculation, short-term memory, language comprehension, spatial awareness, and ability to perform tasks. The assessment typically takes 5 to 10 minutes to administer. The maximum score is 30 points, with higher scores indicating better cognitive abilities. Each correct answer earns one point. A total score of <= 24 indicates mild cognitive impairment, while a score below 16 indicates severe cognitive impairment (Bleecker, Bolla-Wilson, Kawas, & Agnew, 1988). However, these cutoffs should be adjusted according to educational level: for individuals with elementary education or less, <= 20 indicates mild cognitive impairment, and <= 16 indicates severe cognitive impairment.
Geriatric depression assessment (GDS) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Geriatric Depression Scale assesses 15 items reflecting the individual's condition over the past week. Points are assigned as follows: Questions 1, 5, 7, 11, and 13 score 1 point if answered "No"; Questions 2, 3, 4, 6, 8, 9, 10, 12, 14, and 15 score 1 point if answered "Yes". Data is obtained through observation, interviews with the individual or caregivers. The total score ranges from 0 to 15 points. Cutoff points: Scores of 0-4 indicate good mental and emotional adaptation. Scores of 5-9 suggest mild depressive tendencies, recommending psychological counseling or professional consultation. Scores of 10-15 indicate more severe depressive tendencies, recommending referral to psychiatric treatment or professional counseling.
Functional oral intake assessment (FOIS) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Functional Oral Intake Assessment consists of 7 items used to evaluate and observe how individuals consume food and liquids orally, categorized into stages 1-7. Stage 1 indicates no oral intake, while stage 7 indicates unrestricted oral intake with no limitations. The assessment is based on observing the individual's eating and swallowing abilities or reviewing institutional dietary records. Cutoff points: Stages 1-3 indicate dependence on tube feeding, while stages 4-7 indicate full oral intake.
Difficulty of mouth process (DOMP) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Swallowing Difficulty Index is used to observe the severity of swallowing difficulties in study subjects, categorized into 0-4 stages. Stage 0 indicates severe difficulty, with significant oral residue, food scattered to the cheeks and beside the tongue, and frequent drooling. Stage 2 indicates moderate severity, with slow eating speed, poor water flow dynamics, some residue beside the tongue, and possible drooling. Stage 3 indicates mild severity, with slightly slower eating speed, slightly open lips, and occasional drooling. Stage 4 indicates normal swallowing function.
Oral health assessment tool (OHAT) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Oral Health Assessment Scale consists of 8 assessment items: lips, tongue, gums, toothache, saliva, teeth, dentures, and oral hygiene. Each item is scored from 0 to 2 points, where 0 points indicate health and 2 points indicate poor health. Higher scores indicate worse oral health. Data is collected by assessing the individual's oral condition or checking institutional records.
  Score calculation: Scores range from 0 to 16 points, with higher scores indicating poorer oral health.
Swallowing-related quality of life assessment (SWQOL) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The Swallowing Quality of Life Questionnaire consists of 9 assessment items totaling 40 questions and 5 situational inquiries. It assesses the individual's experiences over the past month, their perception of their swallowing ability, and their sensations during swallowing.
  Scoring criteria: Items 1-9 (total of 40 questions) are scored on a 5-point Likert scale: "Always" scores 1 point (90-100% frequency/intensity), "Often" scores 2 points (60-80% frequency/intensity), "Sometimes" scores 3 points (30-50% frequency/intensity), "Rarely" scores 4 points (10-20% frequency/intensity), and "Never" scores 5 points (0% frequency/intensity). Questions 10-14 are supplemented by situational inquiries.Score calculation: Scores range from 40 to 200 points, with higher scores indicating better daily functioning and better quality of life.
Iowa Oral Performance Instrument (IOPI) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  IOPI was used to measure tongue strength, tongue endurance, tongue endurance time, saliva swallowing pressure, effortful saliva swallowing pressure, and the strength of the left and right lips.
Mini-nutrition assessment(MNA) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  To assess the nutritional status of elderly individuals, the scale consists of a total of 18 items divided into nutritional screening (total score of 14 points) and general assessment (total score of 16 points), resulting in a maximum total score of 30 points. Each item is graded according to its scoring level.
  If the nutritional screening score is 11 or less, further nutritional assessment is required, completing questions G-R to determine the "malnutrition indicator value." Nutritional assessment: Complete assessments for questions G-R, incorporate them into the total assessment score, and determine the "malnutrition indicator value." Cutoff points: 24 to 30 points = normal nutritional status; 17 to 23.5 points = at risk of malnutrition; less than 17 points = malnourished.
Repetitive saliva swallowing test (RSST) | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  The repetitive saliva swallowing test measures the number of rapid swallows in 30 seconds. The difficulty swallowing index during the pharyngeal phase will be used to observe the number of times the individual swallows saliva in 30 seconds, with a total of 3 assessment items. 1 point is scored if it does not reach three times, and 0 points are scored if the sensation of swallowing motion cannot be felt on the Adam's apple. The cutoff points are as follows: a score of 1 or below indicates a high-risk group for chewing and swallowing disorders, while a score of 2 indicates normal swallowing function.
Aspiration assessment | T1 baseline; Outcomes were measured 6 times, T2~T7 were conducted at 4.8.12.24.36.48 weeks after exercise.
  To obtain information for each option, use the aspiration assessment form to interview the case or caregiver, or check the institution's records: whether there has been a physician-diagnosed pneumonia, fever ≥ 38℃, respiratory symptoms like coughing or difficulty breathing, and the dates of occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Kao S Hua, Master, Study Chair — Chang Gung Memorial Hospital at Linkou, Taipei Medical University, Taipei, Taiwan
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan, Taoyuan City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Jones E, Speyer R, Kertscher B, Denman D, Swan K, Cordier R. Health-Related Quality of Life and Oropharyngeal Dysphagia: A Systematic Review. Dysphagia. 2018 Apr;33(2):141-172. doi: 10.1007/s00455-017-9844-9. Epub 2017 Sep 2. PMID 28866854
- [Background] Lazarus C, Logemann JA, Huang CF, Rademaker AW. Effects of two types of tongue strengthening exercises in young normals. Folia Phoniatr Logop. 2003 Jul-Aug;55(4):199-205. doi: 10.1159/000071019. PMID 12802092
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Park T, Kim Y. Effects of tongue pressing effortful swallow in older healthy individuals. Arch Gerontol Geriatr. 2016 Sep-Oct;66:127-33. doi: 10.1016/j.archger.2016.05.009. Epub 2016 Jun 3. PMID 27318884
- [Background] Rech RS, de Goulart BNG, Dos Santos KW, Marcolino MAZ, Hilgert JB. Frequency and associated factors for swallowing impairment in community-dwelling older persons: a systematic review and meta-analysis. Aging Clin Exp Res. 2022 Dec;34(12):2945-2961. doi: 10.1007/s40520-022-02258-x. Epub 2022 Oct 7. PMID 36207669
- [Background] Robbins J, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, Taylor AJ. The effects of lingual exercise in stroke patients with dysphagia. Arch Phys Med Rehabil. 2007 Feb;88(2):150-8. doi: 10.1016/j.apmr.2006.11.002. PMID 17270511
- [Background] Sakai K, Nakayama E, Yoneoka D, Sakata N, Iijima K, Tanaka T, Hayashi K, Sakuma K, Hoshino E. Association of Oral Function and Dysphagia with Frailty and Sarcopenia in Community-Dwelling Older Adults: A Systematic Review and Meta-Analysis. Cells. 2022 Jul 14;11(14):2199. doi: 10.3390/cells11142199. PMID 35883642
- [Derived] Kao SH, Chu H, Banda KJ, Sung CM, Chen R, Chang LF, Chiang KJ, Pien LC, Chou KR. Effects of Tongue Resistance and Strengthening Exercises on Tongue Strength and Oropharyngeal Swallowing in Frail Older Adults With Mild Cognitive Impairment: A Double-Blind Randomised Controlled Trial. J Oral Rehabil. 2026 Feb;53(2):402-414. doi: 10.1111/joor.70087. Epub 2025 Nov 5. PMID 41190776